CLINICAL TRIAL: NCT05031208
Title: Research on the Acute and Long Term Effects on Memory and the Mechanism of Action of Vagus Nerve Stimulation in Patients With Refractory Epilepsy
Brief Title: Acute and Long Term Effects of VNS on Memory in Patients With Refractory Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: EC/2016/0786
Record Dates: First submitted 2021-08-19; First posted 2021-09-01 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Refractory Epilepsy
Keywords: Vagus nerve stimulation; Transcutaneous vagus nerve stimulation; Word recognition paradigm
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vagus nerve stimulation (Experimental): Invasive vagus nerve stimulation
  Interventions: Diagnostic Test: Memory task
- Transcutaneous vagus nerve stimulation (Experimental): Cymba concha stimulation
  Interventions: Diagnostic Test: Memory task
- Sham vagus nerve stimulation (Sham Comparator): No vagus nerve stimulation
  Interventions: Diagnostic Test: Memory task

INTERVENTIONS:
Diagnostic Test: Memory task — Word recognition task

SUMMARY:
Refractory epilepsy patients implanted with a vagus nerve stimulator perform a memory test at baseline in three conditions: invasive vagus nerve stimulation (VNS), transcutaneous vagus nerve stimulation (taVNS) and sham stimulation. After 6 weeks of VNS treatment, the memory test is repeated in two condition: invasive vagus nerve stimulation (VNS) and sham stimulation.

The endpoint of this experiment is assessing the effect of VNS and taVNS on memory performance.

DETAILED DESCRIPTION:
Previous studies underlined the potential of both invasive as transcutaneous auricular vagus nerve stimulation to ameliorate certain cognitive functions.

In this randomized, controlled cross-over within-subjects study, a memory test is conducted in patients with refractory epilepsy who are implanted with a vagus nerve stimulation.

The memory test consists out of a word recognition paradigm based on the study of Clarck et al. published in 1999 in Nature Neuroscience. Testing is performed at baseline (before start of the stimulation) and after 6 weeks of treatment with vagus nerve stimulation.

During the first session, the patients complete the word recognition task during three interventions:

* Invasive vagus nerve stimulation
* Transcutaneous vagus nerve stimulation (cymba concha)
* Sham vagus nerve stimulation (no stimulation)

During the second session, the patients complete the word recognition task during two interventions:

* Invasive vagus nerve stimulation
* Sham vagus nerve stimulation (no stimulation)

The goal is to investigate if invasive vagus nerve stimulation and transcutaneous nerve stimulation can influence (i.e. improve) the performance on the memory task and if this performance is improved after 6 weeks of VNS treatment.

ELIGIBILITY:
Inclusion Criteria:

* Refractory epilepsy
* Treated with vagus nerve stimulation
* IQ >= 70 and able to perform the memory task

Exclusion Criteria:

* IQ < 70

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-11-22 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2020-08-28 (Actual)

PRIMARY OUTCOMES:
Immediate recall score at session 1 | At baseline
  Free recall score for correctly recalled words (min score 0,max score 21, higher score indicates better performance), calculated as a percentage
Immediate recall score at session 2 | After 6 weeks of VNS treatment
  Free recall score for correctly recalled words (min score 0, max score 21, higher score indicates better performance)), calculated as a percentage
Delayed recognition scores at session 1 | At baseline
  Hitscore for correctly recognized target words (min score 0,max score 63, higher score indicates better performance), score for not recognized target words= misses (min score 0,max score 63, higher score indicates worse performance),correct rejection score of non-target related words (min score 0,max score 63, higher score indicates better performance), score for incorrect recognition of non-target related words= false alarms (min score 0,max score 63, higher score indicates worse performance), discrimination index= hit score -false alarm score (min score 0,max score 63, higher score indicates better performance). All scores are calculated as a percentage.
Delayed recognition scores at session 2 | After 6 weeks of VNS treatment
  Hitscore for correctly recognized target words (min score 0,max score 48, higher score indicates better performance), score for not recognized target words= misses (min score 0,max score 48, higher score indicates worse performance),correct rejection score of non-target related words (min score 0,max score 48, higher score indicates better performance), score for incorrect recognition of non-target related words= false alarms (min score 0,max score 48, higher score indicates worse performance), discrimination index= hit score -false alarm score (min score 0,max score 48, higher score indicates better performance). All scores are calculated as a percentage.

SECONDARY OUTCOMES:
Attention score at session 1 | At baseline
  Score of correct responses on 6 open question (min score 0, max score 6, higher score indicates better performance), calculated as a percentage
Attention score at session 2 | After 6 weeks of VNS treatment
  Score of correct responses on 6 open question (min score 0, max score 6, higher score indicates better performance), calculated as a percentage

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Clark KB, Naritoku DK, Smith DC, Browning RA, Jensen RA. Enhanced recognition memory following vagus nerve stimulation in human subjects. Nat Neurosci. 1999 Jan;2(1):94-8. doi: 10.1038/4600. PMID 10195186
- [Background] Jacobs HI, Riphagen JM, Razat CM, Wiese S, Sack AT. Transcutaneous vagus nerve stimulation boosts associative memory in older individuals. Neurobiol Aging. 2015 May;36(5):1860-7. doi: 10.1016/j.neurobiolaging.2015.02.023. Epub 2015 Feb 28. PMID 25805212
- [Background] Colzato LS, Ritter SM, Steenbergen L. Transcutaneous vagus nerve stimulation (tVNS) enhances divergent thinking. Neuropsychologia. 2018 Mar;111:72-76. doi: 10.1016/j.neuropsychologia.2018.01.003. Epub 2018 Jan 8. PMID 29326067
- [Background] Steenbergen L, Sellaro R, Stock AK, Verkuil B, Beste C, Colzato LS. RETRACTED: Transcutaneous vagus nerve stimulation (tVNS) enhances response selection during action cascading processes. Eur Neuropsychopharmacol. 2015 Jun;25(6):773-8. doi: 10.1016/j.euroneuro.2015.03.015. Epub 2015 Mar 30. PMID 25869158
- [Derived] Mertens A, Gadeyne S, Lescrauwaet E, Carrette E, Meurs A, De Herdt V, Dewaele F, Raedt R, Miatton M, Boon P, Vonck K. The potential of invasive and non-invasive vagus nerve stimulation to improve verbal memory performance in epilepsy patients. Sci Rep. 2022 Feb 7;12(1):1984. doi: 10.1038/s41598-022-05842-3. PMID 35132096